CLINICAL TRIAL: NCT02747589
Title: Study to Assess the Feasibility of Stimulating the Visual Cortex in Blind Volunteers
Brief Title: Feasibility of Stimulating the Visual Cortex in Blind
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ausaf A. Bari, MD, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BlindStim
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Blindness,Acquired
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Subjects will be implanted to assess the feasibility of stimulating visual cortex to restore vision in blind volunteers.
  Interventions: Procedure: Surgical device implant in brain

INTERVENTIONS:
Procedure: Surgical device implant in brain — Neuropace RNS implant ove visual cortex

SUMMARY:
In this study, the investigators intend to evaluate the use of a commercially available neurostimulator system, NeuroPace RNS System to stimulate the visual cortex. The NeuroPace RNS System has a proven record of safety and reliability was approved by the FDA in November 2013. The RNS System is indicated for use in patients with epilepsy and includes a skull implanted neurostimulator. No modification to the RNS System is required for this study. This study will use this device to better understand the effect of stimulation on the visual parts of the brain.

The main purposes of this study are to confirm the desired location to implant a device in the visual cortex, determine the amount of energy needed to elicit vision, and assess the nature of the vision that is produced. This information is important to have early in the process of designing a visual cortical prosthesis that could eventually be used for commercial use.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is blind (i.e. bare light perception or no light perception in both eyes).
2. Subject has a history of useful form vision.
3. Subject is between the age of 18-74.
4. Subject resides within 2 hours distance (by ground transportation) of the investigational site.
5. Subject is (a) male or (b) a female of childbearing potential with a negative pregnancy test who is using a reliable method of contraception or is at least two years post-menopause.
6. Subject is able to complete regular office and telephone appointments per the protocol requirements.
7. Subject is medically fit for neurosurgical intervention.
8. Subject is considered a good candidate to be implanted with the investigational device.

Exclusion Criteria:

1. Subject is blind due to cortical etiology (e.g. injury to the visual cortex).
2. Subject is eligible for another commercially available vision restoration therapy (e.g. retinal prosthesis).
3. Subject is at high risk for surgical complications such as active systemic infection, coagulation disorders (such as the use of anti-thrombotic therapies) or platelet count below 100,000.
4. Subject has history of bleeding or immune compromise.
5. Subject is taking chronic anticoagulants or antiplatelet agent or subject has an abnormally elevated preoperative coagulation profile (either PTT or PT/INR).
6. Subject has had prior craniotomy or brain surgery.
7. Subject has evidence of active intracranial disease that would preclude elective neurosurgical intervention, such as unruptured intracranial aneurysm or brain tumor, or aberrant visual cortex anatomy, such as prior stroke or arteriovenous malformation.
8. Subject has a significant abnormality on preoperative brain MRI
9. Subject has a prior history of seizures or epilepsy.
10. Subject has Parkinson's disease
11. Subject has a prior history of serious head injury with loss of consciousness.
12. Subject has a progressive central nervous system disease.
13. Subject has history of implant-related infection.
14. Implantation of the investigational device would present unacceptable risk.
15. Subject requires or is likely to require any of the following medical procedures while implanted with the NeuroPace RNS System: MR imaging, diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS). These medical procedures are contraindicated for patients with an implanted RNS® System. Energy from these procedures can be sent through the implanted brain stimulation system and cause permanent brain damage which may cause severe injury, coma, or death. Brain damage can occur from any of the listed procedures even if the RNS® Neurostimulator is turned off or if the Leads are not connected to the Neurostimulator, and can occur even if the Neurostimulator has been removed and any Leads (or any part of a Lead) or the cranial prosthesis remain. Refer to the Contraindications section of the RNS System User Manual for further details.
16. Subject is implanted with any neurostimulation or neuromodulation device in the head including, but not limited to cochlear implant, deep brain stimulator, or auditory brain implant.
17. Subject has a clinically significant or unstable medical condition including uncontrolled systemic hypertension with values above 170/100; cardiac or pulmonary disease; uncorrected coagulation abnormalities; diabetes; or any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.
18. Subject has had an alcohol or illicit substance use disorder within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response.
19. Subject has uncontrolled chronic pain.
20. Subject has significant neurocognitive impairment in memory domain (based on MoCA-BLIND <18 or WAIS-IV <80, described below).
21. Subject had moderate or severe depression, as determined by a score of at least 17 on the HAMD.
22. Subject has had a suicide attempt in the last two years, presence of a suicide plan (an answer of "Yes" to Question C4 in Section C-Suicidality of MINI International Neuropsychiatric Interview), or a "yes" answer to any one of the ten suicidal ideation and behavior questions on the C-SSRS.
23. Subject has a disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

    1. Cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease
    2. Psychiatric disease including diagnosed forms of depression
    3. Does not speak a principal language associated with the region
    4. Deafness or selective frequency hearing loss that prevents adequate communication with the researchers.
24. Subject is pregnant or planning on becoming pregnant in the next year.
25. Subject is enrolled in another therapeutic investigational drug or device trial

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stimulation level required to elicit visual phosphene | 6 months
  Quantitative outcome. Direct brain stimulation to reproduce visual phenomena has not been done. There are no predesigned outcome measures. For this outcome measure, we will determine how much stimulation (in amps) is required to induce a perception of vision.
Characterization of stimulation-induced visions | 6 months
  Descriptive outcome. Subjects will be asked to describe the type of visual perception that is induced by direct brain stimulation.
Spatial localization of stimulation to produce visual phenomena with direct cortical stimulation. | 6 months
  Anatomic outcome. No predetermined outcome scale exists. We will assess patients and the sites of brain stimulation to determine which areas of the brain produce reliable visual phenomena when stimulated.

CONTACTS AND LOCATIONS:
Overall Officials: Ausaf Bari, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Neurosurgery, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No